CLINICAL TRIAL: NCT01274754
Title: Perioperative Administration of Erythromycin and Brain Protection
Brief Title: Neuroprotection With Erythromycin in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Evanthia Thomaidou, Consultant Anesthesiologist, AHEPA University Hospital
Other Study IDs: VRTE
Record Dates: First submitted 2010-03-01; First posted 2011-01-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Functional Disturbances Following Cardiac Surgery
Keywords: neuroprotection; erythromycin; neurocognitive assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken from all patients for the detection of tau protein, IL-1 and IL-6,
  1. preoperatively
  2. 12 hours after surgery
  3. the 6th day after surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- erythromycin group: Patients of erythromycin group: 25mg/kg erythromycin intravenously 12 hours before surgery and 12 hours after the end of surgery.
- control group: no administration of erythromycin

SUMMARY:
Neurological complications occur in open heart surgery with a frequency of 40% and they range from major neurological deficits (due to a stroke) to neurocognitive and behavioral disorders. This study aims to determine if erythromycin, a worldwide known antibiotic, protects the brain from damage when given in high doses before and during open heart surgery.

The investigators consume that high dose of erythromycin will protect the brain with a pharmacological preconditioning against the global ischemia during the perioperative period of heart surgery.

DETAILED DESCRIPTION:
First Version: Study Protocol Authors: Thomaidou E., Vretzakis G., Argiriadou E., Stamatiou G., et al.

Perioperative administration of erythromycin and brain protection

Study Setting: On-pump, planned cardiac surgery. Randomized, double blinded clinical trial of two parallel groups. Group A: control group. Group B: erythromycin group (dose 25mg/kg intravenously).

Purpose:

Neurological complications occur in open heart surgery with a frequency of 40% and they range from major neurological deficits (due to a stroke) to neurocognitive and behavioral disorders. This study aims to determine if erythromycin, a worldwide known antibiotic, protects the brain from damage when given in high doses before and during open heart surgery.

Hypothesis:

The investigators consume that high dose of erythromycin will protect the brain with a pharmacological preconditioning against the global ischemia during the perioperative period of heart surgery.

The aims of this study are:

1. To determine the effect of high-dose perioperative erythromycin administration on neurological outcome in patients undergoing cardiac surgery
2. To determine the relationship of neurological monitoring, specifically NIRS, to neurological outcomes and to determine if erythromycin affects this relationship.

Preoperative Period

Patient Exclusion Criteria: patients > 80 years old, cerebrovascular disease with residual deficits, stroke, alcoholism, psychiatric disease.

Preoperative patient neurocognitive status assessment from the same clinical psychologist in all patients:

at least one day before surgery, perform neurocognitive tests.

Patients of group A: 25mg/kg erythromycin intravenously 12 hours before surgery.

Intraoperative Period

Cerebral monitoring: continuous measurement and registration of cerebral oximetry data (NIRS - INVOS), record of frequency and duration of desaturation episodes (a fall >20% compared to baseline values) and record of interventions to correct desaturation.

Anaesthesia depth monitoring: continuous measurement of bispectral index (BIS).

Registration of: duration of CPB and cross clamp time, mean arterial pressure, heart rate, temperature and ETCO2.

Anesthesia Procedures: anesthesia induction with fentanyl 10-15μg/kg, propofol 2gm/kg and rocuronium 0,6mg/kg. Anesthesia maintenance with propofol.

Postoperative Period - ICU

Postoperative patient neurocognitive status assessment from the same clinical psychologist in all patients:

On discharge, and 3 months later perform neurocognitive tests.

Patients of group A: will receive high dose of erythromycin 12 hours after the end of surgery.

Registration of:

Post operative blood loss, duration of ICU stay, mechanical ventilation duration, duration of hospital stay, inotropic support, postoperative myocardial infarction, re-operation, dialysis, neurocognitive decline, other complications.

BIOCHEMICAL INDEX

Blood samples will be taken from all patients for the detection of tau protein, IL-1 and IL-6,

1. preoperatively
2. 12 hours after surgery
3. the 6th day after surgery

ELIGIBILITY:
Inclusion Criteria:

* patients < 80 years old scheduled for elective cardiac surgery coronary artery bypass grafting, good cooperation with the clinical psychologist

Exclusion Criteria:

* patients > 80 years old
* cerebrovascular disease with residual deficits
* stroke
* alcoholism
* psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective cardiac surgey coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
biochemical markers of brain ischemia and intraoperative cerebral oxymetry data | September 2010

SECONDARY OUTCOMES:
better neurocognitive outcome in Erythromycin group | November 2010

CONTACTS AND LOCATIONS:
Overall Officials: George Vretzakis, Prof., Study Director — University of Thessaly
Locations (2):
- Greece (2):
  - Ahepa University Hospital, Thessaloniki, Hotmail
  - Ahepa University Hospital, Thessaloniki

REFERENCES:
- [Derived] Thomaidou E, Argiriadou H, Vretzakis G, Megari K, Taskos N, Chatzigeorgiou G, Anastasiadis K. Perioperative Use of Erythromycin Reduces Cognitive Decline After Coronary Artery Bypass Grafting Surgery: A Pilot Study. Clin Neuropharmacol. 2017 Sep/Oct;40(5):195-200. doi: 10.1097/WNF.0000000000000238. PMID 28816833